CLINICAL TRIAL: NCT02173327
Title: Continuously Helm CPAP Versus Intermittent Mask CPAP After Major Abdominal Surgery
Brief Title: Helm CPAP Versus Mask CPAP After Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Klaus Vennick Marcussen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHPOTA-01
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuously Helm CPAP (Other): Continuously helm CPAP for 6 hours
  Interventions: Device: Continuously helm CPAP
- Intermittent Mask CPAP (Other): Intermittent Mask CPAP for 10minuttes every 2 hours in a 18 hours period postoperative.
  Interventions: Device: Intermittent Mask CPAP

INTERVENTIONS:
Device: Continuously helm CPAP — 6 hours
  Arms: Continuously Helm CPAP
Device: Intermittent Mask CPAP — 10min every 2 hour for 18 hours
  Arms: Intermittent Mask CPAP

SUMMARY:
Postoperative pulmonal complications (Abbreviation - PPC) after major abdominal surgery remains a significant clinical problem delaying rehabilitation after surgery. CPAP is one approach to minimize the frequency and severeness of PPC.

In the investigators' organization intermittent mask CPAP every 2 hour, 15min, is used routineously after major abdominal surgery.

Recently new devices has been designed, which give the opportunity tip deliver continuously CPAP with out interruptions because of presumed better comfort. Therefore better patient compliance.

No studies to date have investigated the possible benefit of using continuously helm CPAP versus the traditional intermittent mask CPAP after major abdominal surgery.

The investigators' study will investigate if there are any benefits with continuously Helm CPAP Versus intermittent Mask CPAP After Major Abdominal Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective major abdominal surgery

Exclusion Criteria:

* Severe lung disease. Airway deformity. Need for CPAP at home. Ongoing oxygen therapy. Cannot give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 | 24 hours
  Measured 6,12 and 18 hours after surgery

SECONDARY OUTCOMES:
V/Q mismatch | 24 hours
  V/Q mismatch measured with ALPE essential®. Meassured preoperative, on arrival in the postoperative ward and 24 hours postoperative.
Postoperative complications | 30 days
  Pulmonal complications defined as; needs of oxygen therapy more than 3 days after surgery, pneumonia and x-ray verified atelektases within 30 days after surgery.
Length of stay | 30 days
  Length of stay
Admittance to the intensive care unit | 30 days
  If needed. Cause and length of stay in the intensive care unit i recorded.
Mortality | 30 days
  Mortality

OTHER OUTCOMES:
Total CPAP therapy time | 24 timer
  Measured in total minutes
CPAP interruptions | 24 timer
  Length and cause of the interruptions are noted
Comfort during CPAP therapy | 24 timer
  The comfort during CPAP therapy. Measured on an numeric rang scale from 0-10, where 0 is no discomfort and 10 is extensive discomfort during CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Christian R Mortensen, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Osterkamp JTF, Strandby RB, Henningsen L, Marcussen KV, Thomsen T, Mortensen CR, Achiam MP, Jans O. Comparing the effects of continuous positive airway pressure via mask or helmet interface on oxygenation and pulmonary complications after major abdominal surgery: a randomized trial. J Clin Monit Comput. 2023 Feb;37(1):63-70. doi: 10.1007/s10877-022-00857-7. Epub 2022 Apr 16. PMID 35429325